CLINICAL TRIAL: NCT06884566
Title: Effect of Acute Supplementation (taurine) on Maximal Strength and Anaerobic Power
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Lancashire Cyprus (Other)
Responsible Party: Principal Investigator, Kyriaki Antoniou, Associate Lecturer, University of Central Lancashire Cyprus
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: ΕΕΒΚ/ΕΠ/2024/76
Record Dates: First submitted 2025-01-23; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-01

CONDITIONS: Taurine
Keywords: Taurine; Power; Strenght; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Taurine supplementation (Experimental): Participants consumed 50mg·kg -1 of taurine diluted in 500ml of a sugar-free lemonade drink.
  Interventions: Dietary Supplement: Taurine supplementation
- Placebo (Placebo Comparator): Placebo was a 500ml sugar-free lemonade drink with nothing added
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Taurine supplementation — For the intervention trials participants consumed the following in randomized order: 50mg·kg -1 of taurine diluted in 500ml of a sugar-free lemonade drink or placebo which was a sugar-free lemonade drink with nothing added, 60 minutes before the exercise protocols. Participants wore a nose plug during consumption to confirm that no taste differences were discernible between trials.
  Arms: Taurine supplementation
Dietary Supplement: Placebo — For the intervention trials participants consumed the following in randomized order: 50mg·kg -1 of taurine diluted in 500ml of a sugar-free lemonade drink or placebo which was a sugar-free lemonade drink with nothing added, 60 minutes before the exercise protocols. Participants wore a nose plug during consumption to confirm that no taste differences were discernible between trials.
  Arms: Placebo

SUMMARY:
This crossover-design study examines the acute effect of taurine on trained individuals aged 18-40 on strength and power outputs.

DETAILED DESCRIPTION:
The purpose of this study is to further investigate any potential ergogenic effects offered by taurine, under specific conditions, namely that of acute supplementation, as opposed to the chronic supplementation protocols of many popular ergogenic aids, such as creatine and beta alanine. Exercise modes investigated include maximal isometric strength, maximal instantaneous power generation, and sustained maximal anaerobic power output, investigated via grip strength, vertical jump height, and the Wingate test, respectively.

ELIGIBILITY:
Inclusion Criteria:

* participants 18 - 40 years of age
* physically active or recreationally active with consistent training more than 3 times per week for at least 6 months
* non-smokers

Exclusion Criteria:

* cardiovascular, respiratory or metabolic diseases
* any musculoskeletal injury in the last six months
* taking taurine and/or creatine supplementation in the past three months

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Maximal Isometric strength in kilograms assessed via handgrip test | Day 1
Relative Isometric strength in kilograms assessed via handgrip test | Day 1
Maximal Instantaneous power generation in W/kg assessed via vertical jump height test. | Day 1
Average Instantaneous power generation in W/kg assessed via vertical jump height test. | Day 1
Peak power in Watts assessed via the Wingate Anaerobic test | Day 1
Maximal Isometric strength in kilograms assessed via handgrip test | After 48 hours
Relative Isometric strength in kilograms assessed via handgrip test | After 48 hours
Maximal Instantaneous power generation in W/kg assessed via vertical jump height test. | After 48 hours
Average Instantaneous power generation in W/kg assessed via vertical jump height test. | After 48 hours
Peak power in Watts assessed via the Wingate Anaerobic test | After 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Efstathios Christodoulides, PhD, Principal Investigator — https://www.uclancyprus.ac.cy/
Locations (1):
- University of Central Lancashire Cyprus, Larnaca, Pyla, Cyprus

IPD SHARING:
Plan to Share IPD: No